CLINICAL TRIAL: NCT04395651
Title: The Role of 18F-FDG-PET/CT Scan in Lung Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Walaa Otify Thabet, Assistant Lecturer-principal investigator, Assiut University
Other Study IDs: PET/CT in lung cancer
Record Dates: First submitted 2020-05-13; First posted 2020-05-20 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: PET/CT — It is a prospective clinical study that will include patients known to have lung cancer and referred to nuclear medicine unit to perform 18F-FDG PET/CT for staging and therapy planning as well as patients referred for assessment of response of therapy and restaging.

SUMMARY:
Describe strengths and limitations of FDG PET/CT for staging. Evaluate the utility of PET/CT in assessment of therapy response and restaging

DETAILED DESCRIPTION:
Lung cancer is one of the most common cancers and it represents the main cause of cancer mortality worldwide.

It is histopathological classified into main groups: Small cell lung cancer (15%) and Non-small cell lung cancer (85%). NSCLCs are generally subcategorized into adenocarcinoma, squamous cell carcinoma (SqCC), and large cell carcinoma. Positron emission tomography (PET) is now an important cancer imaging tool, both for diagnosis and staging, as well as offering prognostic information based on response.

PET sets the gold standard in the evaluation of an indeterminate solitary pulmonary nodule or mass, where PET has proven to be significantly more accurate than computed tomography (CT).

For NSCLC chest CT is the standard imaging modality for assessing primary tumor size and identifying its margins. PET-CT may be helpful in assessing a nodule located in same lobe. It can also provide information on parietal or mediastinal involvement. PET is useful for differentiating tumor tissue from atelectasis, which may be helpful if radiotherapy is planned to determine the target volume .

In the evaluation of metastatic spread to loco-regional lymph nodes, PET is significantly more accurate than CT, so that invasive surgical staging may be omitted in many patients with negative mediastinal PET images.

In patients with positive mediastinal PET images, invasive surgical staging remains mandatory because of the possibility of false-positive findings due to inflammatory nodes or granulomatous disorders.

Forty percent of patients with NSCLC have distant metastases at presentation, most commonly in the adrenal glands, bones, liver, or brain .

In the search for metastatic spread, PET is a useful adjunct to conventional imaging. This may be due to the finding of unexpected metastatic lesions or due to exclusion of malignancy in lesions that are equivocal on standard imaging. However, at this time, PET does not replace conventional imaging.

The diagnostic accuracy of initial pre-therapy PET-CT results in improved staging, and thus is of high prognostic value.

Many studies conducted the value of using semi-quantitative measures as metabolic tumor volume (MTV) and Total lesion glycolysis (TLG) in predicting prognosis and survival rather than the traditional method of measuring Standard uptake value (SUV).

Several studies have demonstrated that PET imaging proves useful for assessing the response to chemo therapy or targeted therapy in patients with metastatic NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically proven lung cancer and referred to nuclear medicine unit to perform PET/CT for staging and patient referred for assessment of response of therapy and re staging.

Exclusion Criteria:

* Pregnant women.
* Patients unable to sleep in a fixed position for 20 minutes.
* Severely ill patients who aren't capable of complying with study procedures or comatose patients.
* Patients with known second primary

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All eligible patients during the period of the study will be included (total coverage).
  Expected number according to patients flow is 30 patients.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
PET/CT in lung cancer | one year
  * Analysis of the number and type of metastatic lesions detected by PET/CT in lung cancer patients(staging).
  * Analysis of the number and type of metastatic lesions detected by PET/CT in lung cancer patients after therapy(re staging).

SECONDARY OUTCOMES:
PET/CT in lung cancer | one year
  -To evaluate risk benefit of PET/CT examination in lung cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Taha Zaky Mahran, Prof.Dr., Study Chair — Assiut University; Ahmad Zaher, Prof .Dr., Study Chair — National Cancer Institute (NCI); Nesreen Mekkawy, Dr., Study Chair — Assiut University

REFERENCES:
- [Background] Ambrosini V, Nicolini S, Caroli P, Nanni C, Massaro A, Marzola MC, Rubello D, Fanti S. PET/CT imaging in different types of lung cancer: an overview. Eur J Radiol. 2012 May;81(5):988-1001. doi: 10.1016/j.ejrad.2011.03.020. Epub 2011 Mar 31. PMID 21458181
- [Background] Huang Y, Liu Z, He L, Chen X, Pan D, Ma Z, Liang C, Tian J, Liang C. Radiomics Signature: A Potential Biomarker for the Prediction of Disease-Free Survival in Early-Stage (I or II) Non-Small Cell Lung Cancer. Radiology. 2016 Dec;281(3):947-957. doi: 10.1148/radiol.2016152234. Epub 2016 Jun 27. PMID 27347764
- [Background] Inamura K. Lung Cancer: Understanding Its Molecular Pathology and the 2015 WHO Classification. Front Oncol. 2017 Aug 28;7:193. doi: 10.3389/fonc.2017.00193. eCollection 2017. PMID 28894699
- [Background] Groheux D, Quere G, Blanc E, Lemarignier C, Vercellino L, de Margerie-Mellon C, Merlet P, Querellou S. FDG PET-CT for solitary pulmonary nodule and lung cancer: Literature review. Diagn Interv Imaging. 2016 Oct;97(10):1003-1017. doi: 10.1016/j.diii.2016.06.020. Epub 2016 Aug 24. PMID 27567555
- [Background] Chao F, Zhang H. PET/CT in the staging of the non-small-cell lung cancer. J Biomed Biotechnol. 2012;2012:783739. doi: 10.1155/2012/783739. Epub 2012 Mar 7. PMID 22577296
- [Background] Quint LE, Tummala S, Brisson LJ, Francis IR, Krupnick AS, Kazerooni EA, Iannettoni MD, Whyte RI, Orringer MB. Distribution of distant metastases from newly diagnosed non-small cell lung cancer. Ann Thorac Surg. 1996 Jul;62(1):246-50. doi: 10.1016/0003-4975(96)00220-2. PMID 8678651
- [Background] Chang CF, Rashtian A, Gould MK. The use and misuse of positron emission tomography in lung cancer evaluation. Clin Chest Med. 2011 Dec;32(4):749-62. doi: 10.1016/j.ccm.2011.08.012. PMID 22054883
- [Background] Ma W, Wang M, Li X, Huang H, Zhu Y, Song X, Dai D, Xu W. Quantitative 18F-FDG PET analysis in survival rate prediction of patients with non-small cell lung cancer. Oncol Lett. 2018 Oct;16(4):4129-4136. doi: 10.3892/ol.2018.9166. Epub 2018 Jul 18. PMID 30214552
- [Background] Yoon DH, Baek S, Choi CM, Lee DH, Suh C, Ryu JS, Moon DH, Lee JS, Kim SW. FDG-PET as a potential tool for selecting patients with advanced non-small cell lung cancer who may be spared maintenance therapy after first-line chemotherapy. Clin Cancer Res. 2011 Aug 1;17(15):5093-100. doi: 10.1158/1078-0432.CCR-10-2791. Epub 2011 Jun 14. PMID 21673067
- [Background] Takahashi R, Hirata H, Tachibana I, Shimosegawa E, Inoue A, Nagatomo I, Takeda Y, Kida H, Goya S, Kijima T, Yoshida M, Kumagai T, Kumanogoh A, Okumura M, Hatazawa J, Kawase I. Early [18F]fluorodeoxyglucose positron emission tomography at two days of gefitinib treatment predicts clinical outcome in patients with adenocarcinoma of the lung. Clin Cancer Res. 2012 Jan 1;18(1):220-8. doi: 10.1158/1078-0432.CCR-11-0868. Epub 2011 Oct 21. PMID 22019513